CLINICAL TRIAL: NCT05528445
Title: Evaluation of Cognitive State in Seniors Using Neurosteer Single-channel EEG With an Auditory Assessment Tool
Brief Title: Evaluation of Cognitive State in Seniors Using Neurosteer EEG System
Status: Completed | Type: Observational
Sponsor: Neurosteer Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 032022
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Decline
Keywords: Cognition; Neurology; EEG; Neurosteer
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients: Patients who are assessed by the clinical staff using Mini-Mental State Exam (MMSE) and Montreal-Cognitive-Assessment-Test(MoCA)
  Interventions: Device: Neurosteer EEG recorder

INTERVENTIONS:
Device: Neurosteer EEG recorder — The system is composed of hardware and software modules that facilitate the capture and interpretation of electrophysiological data as well as enable viewing the processed data in real time and offline. An electrode patch is attached on the subject's forehead to capture the electrophysiological signal. The signal is sent via low energy Bluetooth to an EEG Monitor. The signal is then sent via Wi-Fi to the cloud where the data is stored on a HIPAA compliant server. Data analysis performed in the cloud transforms the electrophysiological signal into easily readable data of brain activity.

SUMMARY:
This is an observational study. Patients who fulfill all inclusion criteria and none of the exclusion criteria will be enrolled in the study, be neurologically evaluated and will go through EEG recordings while listening to an auditory cognitive assessment tool and preforming tasks. EEG recordings will be analyzed using proprietary computational analyses.

DETAILED DESCRIPTION:
One of the major problems in the prevention and treatment of neurological disorders, is the lack of cost effective and reliable tools to assess neurodegeneration on a large scale at a very early stage. Although current imaging methods give a clear image of the brain atrophy involved in neurodegenerative disorders, there are deficiencies prohibiting their usage for prevention-scanning of large high-risk population such as high price, long set-up time and the need for trained personnel to conduct the test. Therefore, the development of a reliable tool to assess brain neurodegeneration, associated with cognitive decline independent of personal interpretation and/or variance between clinicians and between medical facilities would be highly valuable. This tool would allow the healthcare team to make appropriate treatment decisions that could aid in neurodegenerative disease prevention.

The Neurosteer system provides objective neurological biomarkers using a wearable easy-to-use affordable system. The system facilitate the capture and interpretation of EEG data with only a single patch of electrodes, attached on the subject's forehead. Neurosteer examination includes completing auditory tasks while measuring brain activity with the device. The data is analyzed using machine learning methods to produce biomarkers, enabling a report of the patient's activity in real time and offline. The examination is easy to preform and can be conducted in every clinic or in patients' homes.

In this study, clinical staff will identify potential subjects and will examine the eligibility of subject according to inclusion and exclusion criteria. Research staff will inform the patient on study's objective and design. Patients will sign the Informed Consent Form (ICF). Research staff will set up an assessment session using the Neurosteer system. In this session the patient will listen to the auditory assessment battery and perform cognitive tasks. Over the next 7 days, clinical staff will set up another session using the Neurosteer system. In this session the patient will listen to auditory instructions and perform two PASS sub-tasks: a drug sorting task and a phone use task.

Level of cognition will be assessed by validated screening tools (MMSE and MoCA) and the Neurosteer technology.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 50.
* MMSE ≥ 10
* Patient is able to collaborate.
* No seizure events.

Exclusion Criteria:

* Advanced stage of cognitive decline (MMSE < 10).
* Any verbal or non-verbal form of objection from patient or form patient's family member or significant other.
* Significant hearing impairments.
* Significant vision impairments.
* Damage to integrity of scalp and/or skull.
* Skin irritation in the facial and forehead area.
* Epilepsy or seizure activity.
* History of drug abuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients from the inpatient rehabilitation department at Dorot Geriatric Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ady Sasson, Principal Investigator — Dorot, Geriatric Medical Center
Locations (1):
- Dorot - Netanya Geriatric Medical Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molcho L, Maimon NB, Regev-Plotnik N, Rabinowicz S, Intrator N, Sasson A. Single-Channel EEG Features Reveal an Association With Cognitive Decline in Seniors Performing Auditory Cognitive Assessment. Front Aging Neurosci. 2022 May 30;14:773692. doi: 10.3389/fnagi.2022.773692. eCollection 2022. PMID 35707705
- [Background] Maimon NB, Bez M, Drobot D, Molcho L, Intrator N, Kakiashvilli E, Bickel A. Continuous Monitoring of Mental Load During Virtual Simulator Training for Laparoscopic Surgery Reflects Laparoscopic Dexterity: A Comparative Study Using a Novel Wireless Device. Front Neurosci. 2022 Jan 20;15:694010. doi: 10.3389/fnins.2021.694010. eCollection 2021. PMID 35126032
- [Background] Curcic J, Vallejo V, Sorinas J, Sverdlov O, Praestgaard J, Piksa M, Deurinck M, Erdemli G, Bugler M, Tarnanas I, Taptiklis N, Cormack F, Anker R, Masse F, Souillard-Mandar W, Intrator N, Molcho L, Madero E, Bott N, Chambers M, Tamory J, Shulz M, Fernandez G, Simpson W, Robin J, Snaedal JG, Cha JH, Hannesdottir K. Description of the Method for Evaluating Digital Endpoints in Alzheimer Disease Study: Protocol for an Exploratory, Cross-sectional Study. JMIR Res Protoc. 2022 Aug 10;11(8):e35442. doi: 10.2196/35442. PMID 35947423

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients
Started | 77
Completed | 77
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients: Patients who are assessed by the clinical staff using Mini-Mental State Exam (MMSE) and Montreal-Cognitive-Assessment-Test (MoCA)
  Neurosteer EEG recorder: The system is composed of hardware and software modules that facilitate the capture and interpretation of electrophysiological data as well as enable viewing the processed data in real time and offline. An electrode patch is attached on the subject's forehead to capture the electrophysiological signal. The signal is sent via low energy Bluetooth to an EEG Monitor. The signal is then sent via Wi-Fi to the cloud where the data is stored on a HIPAA compliant server. Data analysis performed in the cloud transforms the electrophysiological signal into easily readable data of brain activity.
Arm/Group | Patients
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.28 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 77
MMSE score [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) is a structured assessment tool that evaluates cognitive functioning.
  The MMSE produces a total possible score ranging from 0 to 30. Patients who score below 24 would typically be suspected for cognitive decline or early dementia.
  units on a scale | 26 (4)
MoCA score [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is an assessment tool for the detection of MCI or early dementia. The test assesses the following cognitive domains: visuospatial, naming, memory, attention, language, abstraction, delayed recall and orientation. The scores range from 0 to 30, whereas a score of 26 or above indicates normal cognitive function Population: The number of subjects with a MoCA score is different from the overall number of subjects because some of the subjects were released from the department before undergoing the assessment.
  units on a scale
    number analyzed (Participants) | 58
    (all) | 19.9 (5)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Cognition Level Changes as Evaluated by Current Clinical Tools (i.e. MMSE, MoCA) and Brain Activity Features Extracted Using the Neurosteer Technology.
Description: Cognition level changes will be evaluated by:
  1. Mini Mental State Examination (MMSE). A commonly used assessment tool that evaluates cognitive functioning and produces a total possible score of 30 points. Patients who score below 24 are typically suspected of cognitive decline.
  2. Montreal Cognitive Assessment (MoCA). A commonly used assessment tool that evaluates cognitive functioning. The maximum score is 30, with a score of 26 or higher considered cognitively healthy.
  3. Neurosteer system (single channel EEG recording during cognitive auditory tasks).
  Using data analysis (a variant of the wavelet packet analysis and the best basis algorithm), the EEG signal is transformed into brain activity features (e.g. ST4, A0).
  Pearson correlation will be calculated between the mean activity of the EEG features and individual's MMSE and MoCA scores.
Time Frame: MMSE and MoCA scores will be taken from previous evaluation performed in the institute. Through study completion, brain activity features will be assessed twice within 7 days using the Neurosteer EEG system.
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Patients
Number analyzed (Participants) | 77
Pearson correlation coefficient
  MMSE score + A0 activity | -0.27
  MoCA score + A0 activity | -0.26

ADVERSE EVENTS:
Time Frame: Through study completion, during EEG recordings, up to 1 year.
Description: In this study the risk for any Serious Adverse Events is low, as the nature of the experiment is entirely non-invasive and merely records EEG data.
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT05528445/Prot_SAP_000.pdf